CLINICAL TRIAL: NCT04330456
Title: Combined Treatment of Patients With Soft Tissue Sarcoma Including Preoperative Stereotactic Radiation Therapy and Postoperative Conformal Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SaE in STS
Record Dates: First submitted 2020-03-26; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-02

CONDITIONS: Soft Tissue Sarcoma Adult
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SaE treatment (Experimental): This group will receive combined treatment of soft tissue sarcoma that include 3 steps:
  1. step - preoperative stereotactic radiation therapy in hypofractionation mode (5 fractions 5 Gy each)
  2. step - operation
  3. step - postoperative conformal radiation therapy in normofractionation mode (25 fractions 2 Gy each)
  Interventions: Radiation: Preoperative stereotactic radiation therapy in hypofractionation mode; Procedure: Surgery; Radiation: Postoperative conformal radiation therapy in normofractionation mode

INTERVENTIONS:
Radiation: Preoperative stereotactic radiation therapy in hypofractionation mode — At the first step patient undergoes preoperative stereotactic radiation therapy in hypofractionation mode. Radiation therapy plan is based on topometric MRI and CT scans. Radiation therapy plan are performed after MRI and CT fusion, contouring of the target and surrounding normal tissues.
  At first step only tumor and, if necessary, the surrounding normal tissues, which will be removed during surgery, are exposed to radiation.
  GTV - determined in with the boundaries of the tumor visualised by topometric MRI and CT CTV1 - match GTV CTV2 - formed inward (to the tumor center) from GTV by 0.5-1 cm (depending on the proximity of functionally significant normal tissues (neurovascular bundles, bone tissue, skin and subcutaneous fat, etc.) PTV - 3-5 mm indent from CTV1, taking into account the proximity of functionally significant normal tissues and the planned surgery Preoperative radiation therapy is carried in 5 fractions with a single dose on PTV - 5 Gy, a single dose on CTV2 - 7 Gy.
Procedure: Surgery — In 14-21 days after preoperative stereotactic radiation therapy radical surgery will be performed
Radiation: Postoperative conformal radiation therapy in normofractionation mode — In 25-35 days after the surgery postoperative conformal radiation therapy is performed according to the standard protocol GTV (tumor bed) - based on the volume of the primary tumor, including the swelling zone (T2-weighted images on preoperative MRI) СTV - formed with an indent of 4 cm from GTV (without going beyond the boundaries of the involved compartment), in the transverse direction the indent could be reduced to 2 cm.
  PTV - formed with an indent of 0.5-1cm from CTV An important condition for planning radiation therapy is to limit the dose absorbed during both stages of radiation therapy in surrounding normal tissues that are not removed during surgery.

SUMMARY:
Combined treatment of soft tissue sarcoma includes 3 steps:

1. step - preoperative stereotactic radiation therapy in hypofractionation mode
2. step - operation
3. step - postoperative conformal radiation therapy in normofractionation mode

DETAILED DESCRIPTION:
Combined treatment of soft tissue sarcoma includes 3 steps:

1. At the first step patient undergoes preoperative stereotactic radiation therapy in hypofractionation mode. Radiation therapy plan is based on topometric MRI and CT scans. Radiation therapy plan are performed after MRI and CT fusion, contouring of the target and surrounding normal tissues.

   At first step only tumor and, if necessary, the surrounding normal tissues, which will be removed during surgery, are exposed to radiation.

   GTV - determined in with the boundaries of the tumor visualised by topometric MRI and CT CTV1 - match GTV CTV2 - formed inward (to the tumor center) from GTV by 0.5-1 cm (depending on the proximity of functionally significant normal tissues (neurovascular bundles, bone tissue, skin and subcutaneous fat, etc.) PTV - 3-5 mm indent from CTV1, taking into account the proximity of functionally significant normal tissues and the planned surgery Preoperative radiation therapy is carried in 5 fractions with a single dose on PTV - 5 Gy, a single dose on CTV2 - 7 Gy.
2. Second step is surgery in 14-21 days.
3. In 25-35 days after the surgery postoperative conformal radiation therapy is performed according to the standard protocol GTV (tumor bed) - based on the volume of the primary tumor, including the swelling zone (T2-weighted images on preoperative MRI) СTV - formed with an indent of 4 cm from GTV (without going beyond the boundaries of the involved compartment), in the transverse direction the indent could be reduced to 2 cm.

PTV - formed with an indent of 0.5-1cm from CTV An important condition for planning radiation therapy is to limit the dose absorbed during both stages of radiation therapy in surrounding normal tissues that are not removed during surgery.

ELIGIBILITY:
Inclusion Criteria:

* morphologically verified diagnosis of soft tissue sarcoma
* first diagnosed tumor process
* ability to perform radical surgery
* signed informed consent
* indications for stereotactic and conformal radiation therapy
* no contraindications for radiation and surgical treatment

Exclusion Criteria:

* previous radiation treatment
* acute infection
* pregnancy, lactation
* recurrent tumor
* refuse to sign informed consent
* conditions that can affect the outcome of treatment (immunodeficiency, tuberculosis, etc.)
* tumor topography and volume that don't allow to perform stereotactic and conformal radiation therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Complications | 3 year
  Rate of complications will be measured after completing each step of protocol: stereotactic radiation therapy, surgery and them postoperative conformal radiation therapy

SECONDARY OUTCOMES:
Disease-Free survival | 3 year
  Disease-Free survival will be evaluated after completing the protocol or during the protocol if local recurrence will appear.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center of Oncology named after N.N.Petrov, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No